CLINICAL TRIAL: NCT04664257
Title: Delivering Electronic Cognitive Behavioural Therapy to Patients With Bipolar Disorder and Residual Depressive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Collaborators: Online PsychoTherapy Clinic (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal Investigator, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRY-057-20
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Bipolar Disorder; Bipolar Depression
Keywords: Bipolar Disorder; Bipolar Depression; Cognitive Behavioural Therapy; Virtual Mental Health Care; Psychotherapy
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Randomly assigned to intervention or control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-CBT (Experimental): All e-CBT sessions will be administered through OPTT and will consist of approximately 30 slides per week. The content and format of each weekly online session will be designed to mirror in-person CBT for the treatment of BAD-II. Participants will complete the module and submit the assigned homework to their clinician through OPTT where the clinician will be able to provide personalized feedback. These pre-designed engaging and multimedia modules will be able to streamline the therapy process, helping care providers save time on repeating similar materials to all patients and focusing on delivering personalized feedback to each patient. The slides will highlight a different topic each week and include general information, an overview of skills, and homework that is to be completed within that week. All weekly sessions have an estimated completion time of 50 minutes. During the 12 weeks, both groups will continue with their TAU.
  Interventions: Behavioral: e-CBT
- Treatment as Usual (No Intervention): Participants will continue with treatment as usual and any lifestyle activities (diet, exercise, medication, etc.)

INTERVENTIONS:
Behavioral: e-CBT — e-CBT will be administered with weekly modules. See arm/group descriptions for more information.
  Arms: e-CBT

SUMMARY:
The lifetime prevalence of Bipolar II is 0.4% with the time spent with depressive symptoms outnumbering the time spent with hypomanic symptoms by 35 to 1. Regarding current treatment options, psychotherapy is effective for managing depressive symptoms, with CBT being particularly efficacious. Unfortunately, CBT is often not a feasible treatment option. Electronic CBT (e-CBT) is more accessible for treating various mental illnesses with evidence suggesting it can increase treatment adherence and patient satisfaction. Moreover, e-CBT is suggested to have comparable outcomes to in-person CBT in the treatment of depression and anxiety. Typically, patient-clinician interactions of e-CBT are administered through email however, this is an insecure, unsustainable, and non-scalable treatment delivery method. The proposed study will use the Online Psychotherapy Tool (OPTT), a secure cloud-based platform for the delivery of e-CBT. The aim is to evaluate the feasibility and effectiveness of using OPTT for the treatment of BAD-II with depressive symptoms, while also analyzing social, cultural, and personal factors affecting patients' experience. Participants (n = 80) diagnosed with BAD-II in a depressive episode will be recruited from the Mood and Anxiety Clinic at Providence Care Hospital in Kingston, Ontario, Canada. Eligible participants will then be randomly assigned to either the treatment group (e-CBT plus treatment as usual (TAU)) (n = 40) or the control group (TAU) (n = 40) where they will complete the 12-week program. Participants in the TAU group will be offered the e-CBT program after the first 12 weeks if they wish to take part. Participants in the e-CBT group will complete weekly modules mirroring in-person CBT content and complete homework assignments that will be evaluated by a clinician who will provide personalized feedback through OPTT. Progression/regression of participants will be analyzed using the MADRS, YMRS, and CGI-BP-M questionnaires administered at baseline, after week 6, and after week 12. Personal, social, and cultural factors impacting participant experience will be investigated through an in-depth interview utilizing focus groups. The findings from this study will be the first on the effectiveness of delivering e-CBT to patients with BAD-II with residual depressive symptoms. This approach can provide an innovative method to address the barriers associated with in-person psychotherapy.

DETAILED DESCRIPTION:
Population: Individuals (n = 80) diagnosed with BAD-II who are experiencing an acute depressive episode will be recruited from the Mood and Anxiety Clinic at Providence Care Hospital (PCH) in Kingston, Ontario, Canada. Inclusion criteria include being between 18 and 55 years of age at the start of the study, a confirmed diagnosis of BAD-II according to Diagnostic and Statistical Manual of Mental Health Disorders, 5th Edition (DSM-5), a Montgomery Åsberg Depression Rating Scale (MADRS) score between 7 and 34, competence to consent and participate, the ability to speak and read English, and having consistent and reliable access to the internet. Exclusion criteria include experiencing a current acute hypomanic/manic episode, acute psychosis, severe alcohol or substance use disorder, and active suicidal and/or homicidal ideation. Additionally, if an individual is currently receiving or has received CBT in the past year they will be excluded from the study. To confirm eligibility, participants will undergo a complete assessment from a clinician where the diagnosis will be confirmed using the DSM-5 and a Mini-International National Interview (MINI) version 7.0.2. Eligible participants will be randomly allocated into either the e-CBT plus treatment as usual (TAU) (n = 40) or the control group (TAU exclusively) (n = 40). Participants in the control group will be offered the e-CBT program after the first 12 weeks of the study if they are interested.

Procedure: Upon completion of the initial assessment, if eligible for the study, participants from the e-CBT group will be enrolled in the e-CBT program. All e-CBT sessions will be administered through OPTT and will consist of approximately 30 slides per week. The content and format of each weekly online session will be designed to mirror in-person CBT for the treatment of BAD-II. Participants will complete the module and submit the assigned homework to their clinician through OPTT where the clinician will be able to provide personalized feedback. These pre-designed engaging and multimedia modules will be able to streamline the therapy process, helping care providers save time on repeating similar materials to all patients and focusing on delivering personalized feedback to each patient. The slides will highlight a different topic each week and include general information, an overview of skills, and homework that is to be completed within that week. All weekly sessions have an estimated completion time of 50 minutes. During the 12 weeks, both groups will continue with their TAU. To ensure the quality and consistency of care, care pathways will be fully assigned beforehand, and a clinician will be trained to follow the standard care pathways. Through the training, the clinician will learn the aim and content of each therapeutic session and will be provided with sample homework submissions and modules to better understand how to structure feedback.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar Disorder - 2
* MADRS score of 7-34
* Competence to consent and participate
* Ability to speak and read English
* Consistent and reliable access to the internet

Exclusion Criteria:

* Acute hypomanic/manic episodes
* Acute psychosis
* Severe alcohol or substance use disorder
* Active suicidal and/or homicidal ideation
* Currently receiving/has received CBT in the past year

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms (Montgomery Asberg Depression Rating Scale - MADRS) | Baseline, week 6, week 12
  Clinically validated symptom questionnaire. Scale of 1-6, 6 is worse.
Change in symptoms (Young Mania Rating Scale - YMRS) | Baseline, week 6, week 12
  Clinically validated symptom questionnaire. Scale of 1-4 and 1-8, higher is worse.
Change in symptoms (Modified Clinical Global Impression Scale for Bipolar Disorder - CGI-BP-M) | Baseline, week 6, week 12
  Clinically validated symptom questionnaire. Scale of 1-7 and 1-8, higher is worse.

SECONDARY OUTCOMES:
Differences in personal, social, and cultural factors impacting accessibility to treatment | Week 12 (Post-Treatment)
  Focus groups for providers and patients using Interpretive Phenomenological Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Gutierrez G, Stephenson C, Eadie J, Moghimi E, Omrani M, Groll D, Soares CN, Milev R, Vazquez G, Yang M, Alavi N. Evaluating the Efficacy of Web-Based Cognitive Behavioral Therapy for the Treatment of Patients With Bipolar II Disorder and Residual Depressive Symptoms: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 May 19;12:e46157. doi: 10.2196/46157. PMID 37140460